CLINICAL TRIAL: NCT01968577
Title: Randomized Trial of Creatine-kinase Leak After Rosuvastatin At the Time of Percutaneous Coronary Intervention
Acronym: CLEAR-PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kleber Bomfim Araujo Martins (Other)
Responsible Party: Sponsor-Investigator, Kleber Bomfim Araujo Martins, Doctorate in progress, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBAM-120758
Record Dates: First submitted 2013-10-19; First posted 2013-10-24 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Coronary Artery Disease
Keywords: Coronary angioplasty; Myocardial infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin 40 mg (Experimental): Administration of rosuvastatin 40 mg 2 to 6 hours before percutaneous coronary intervention
  Interventions: Drug: Rosuvastatin
- Control group (No Intervention): The group of patients that do not receive rosuvastatin, 40 mg, before percutaneous coronary intervention.

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 40 mg before percutaneous coronary intervention
  Other Names: Crestor
  Arms: Rosuvastatin 40 mg

SUMMARY:
Patients with stable coronary disease when undergoing percutaneous coronary intervention may present periprocedural myocardial infarction defined at present as a creatine kinase-myocardial isoenzyme (CK-MB) elevation 3 times upper limit of normal, as a cut off for periprocedural myocardial infarction after PCI. Although percutaneous coronary intervention is associated with low rates of complications, periprocedural myocardial infarction has been touted as a negative factor in long-term clinical results . Several clinical, anatomical and technical associate to the occurrence of this event . Although randomized controlled trials and systematic reviews to statin pre intervention have targeted the administration of high-dose statin is recommended before surgery to reduce the risk of periprocedural myocardial infarction, there is no information on the impact of the maximum concentration plasma of statin at the time of percutaneous coronary intervention in stable patients on chronic statin use in preventing periprocedural myocardial infarction or the elevation of cardiac enzymes . The anti-ischemic effect of statins in percutaneous coronary intervention was mainly determined in statin -naïve patients or in patients with acute coronary syndromes . In this work , we studied the impact of the peak plasma concentration of statin at the time of percutaneous coronary intervention was studied through prospective randomized single center in stable patients with chronic statin divided into two groups . In the group (1) Experimental (n = 268 ) was administered at a dose of 40 mg rosuvastatin between one and six hours before surgery and group (2) control without rosuvastatin (n = 268). This range 1 to 6 hours is the time at the peak concentration of rosuvastatin in the blood after oral ingestion. The primary objective was to assess the incidence of periprocedural myocardial infarction by creatine kinase above three times upper normal limit in hospital period and as a secondary objective to analyze the elevation of any amount of creatine kinase on the baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical signs of stable angina (Classification of Canadian Cardiovascular Society 1, 2, 3 or 4) or asymptomatic with evidence of ischemia-induced functional tests with indication of elective PCI.
* Use of statins for a period equal to or greater than 7 days or reported by the patient and confirmed by medical prescription.
* Stent implantation in de novo lesions in native coronary arteries were considered eligible for the study
* The patient or legal representative must sign the consent form before the procedure, in form containing all the details of the research approved by the Ethics Committee of the Institution.

Exclusion Criteria:

* Women of childbearing potential who are not using appropriate contraceptive measures during pregnancy and lactation .
* Values above the upper limit of normal serum levels of CK-MB mass harvested 24 hours prior to the procedure.
* Myocardial infarction < 15 days.
* Renal insufficiency with creatinine clearance < 30 ml/min
* Patients with known allergy, hypersensitivity or contraindication to any of the following: aspirin , heparin , clopidogrel , ticagrelor , and statin or iodinated contrast .
* Participation in other research to influence serum levels of CK-MB mass
* Have taken fibrate 24 hours before the intervention .
* Use of oral anticoagulants or glycoprotein inhibitors at the day of the procedure .
* Evidence of angiographic intracoronary thrombus in the target lesion .
* In -stent restenosis , vein graft or arterial .
* Complications of the procedure as irreversible occlusion of the target vessel as well as branch greater than 1mm in diameter , presence of dissection with compromised flow, caging branch with reduced flow , coronary spasm with abnormal blood flow and distal embolization .
* Inability to deploy stent .
* Use of atherectomy technique .
* Patients were randomized to rosuvastatin be administered prior to the procedure , having the guidewire stent reached the ostium of the coronary target with time less than two hours or having exceeded the period of six hours after oral ingestion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Periprocedural myocardial infarction (Myocardial enzymes arise) | After 12 hours to hospital discharge
  Myocardial enzyme arise 3 times of upper limit of normal, 12 hours of the percutaneous coronary intervention until peak value at hospital discharge.

SECONDARY OUTCOMES:
Any creatine kinase elevation | After 12 hours to hospital discharge
  Any myocardial enzyme arise after 12 hours of the percutaneous coronary intervention until peak value at hospital discharge.

OTHER OUTCOMES:
Hospital mortality | After 12 hours to hospital discharge
  All cause of mortality at the time of the percutaneous coronary intervention to hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Kleber B A Martins, MD, Principal Investigator — Instituto Dante Pazzanese e Cardiologia e Sao Paulo
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo, Brazil